CLINICAL TRIAL: NCT00359736
Title: Vasodilator Therapy and Exercise Tolerance in IPF Patients
Brief Title: Sildenafil Study to Treat Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLIN-009-05F
Record Dates: First submitted 2006-07-31; First posted 2006-08-02 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-09

CONDITIONS: Alveolitis, Fibrosing; Fibrosis, Pulmonary; Hypertension, Pulmonary
Keywords: alveolitis, fibrosing; exercise, aerobic; fibrosis, pulmonary; hypertension, pulmonary
MeSH Terms: conditions — Pulmonary Fibrosis; Hypertension, Pulmonary; Motor Activity | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sildenafil (Experimental): Sildenafil 20 mg tid orally
  Interventions: Drug: sildenafil
- Placebo (Placebo Comparator): Identical Placebo 20 mg tid orally
  Interventions: Drug: sildenafil

INTERVENTIONS:
Drug: sildenafil — Assessing the possible therapeutic benefit of sildenafil on exercise tolerance in IPF patients.
  Other Names: Revatio

SUMMARY:
Medicines that decrease blood pressure in the lungs may help idiopathic pulmonary fibrosis (IPF) patients function better. This study will test whether sildenafil improves the ability to exercise in patients with pulmonary fibrosis of unknown cause.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) is recognized as a predominantly noninflammatory paradigm of lung fibrosis, characterized by heterogeneous myofibroblast proliferation (usual interstitial pneumonia [UIP]) and a poor clinical prognosis. To date no therapies have been demonstrated in well-designed, randomized, controlled trials (RCT) to favorably influence functional status or survival of IPF patients. The need for effective therapies for VA patients with IPF is thus obvious and urgent.

The overall goal of this VA Merit Review clinical research is to generate rigorous preliminary data for evaluation of a new and potentially effective therapy for IPF. The established, combined Miami Veterans Affairs Medical Center (VAMC) - University of Miami (UM) IPF program has participated productively in a number of clinical trials to assess new agents for the therapy of IPF (e.g., interferon gamma-lb, imatinib mesylate, etanercept, bosentan). Our program is uniquely qualified to enroll large numbers of IPF patients in clinical trials, because of its large metropolitan population base (>5,000,000 people) and extensive referral network throughout South and Central America. The Veteran population of South Florida (Dade, Broward and Monroe Counties) is approximately 236,000 (U.S. Census Bureau). Of that number 39% are 65 years of age or older, making them at high risk for IPF. Because of its large Veteran and civilian population base, international referral network and previous experience as a "high enrollment center" in IPF clinical trials, the Miami VAMC-UM IPF program is uniquely qualified to anticipate the role of a CSP lead center.

Our central hypothesis is that sildenafil, a vasodilator, will have a beneficial effect compared to placebo on disease progression, defined as a significant change in the 6-minute walk distance or dyspnea index, in patients with IPF.

Specifically, we will test effects of sildenafil on IPF patients' exercise tolerance and level of dyspnea in a double blind, randomized, placebo controlled (one to one assignment) pilot study. Upon completion of this trial, it will be possible to assess efficacy of sildenafil on progression of disease in IPF and possibly introduce this agent into translational practice. Our specific objectives are:

Specific Objectives 1: To assess the possible therapeutic benefit of a vasodilator, sildenafil, on exercise tolerance in IPF patients.

The working hypothesis is that, compared to placebo, sildenafil will favorably affect rate of decline from baseline in exercise capacity (6-minutes walk).

Specific Objective 2: To assess and compare changes from baseline in pre- and post-exercise dyspnea in sildenafil and placebo control groups.

The working hypothesis is that application of this agent will lead to more sustained exercise and a more favorable clinical outcome in addition to a decrease in the degree of limiting dyspnea after exercise.

The application of vasodilator therapy in IPF is unique in that it directly targets key pathophysiologic mechanisms of functional limitation: Increased pulmonary vascular resistance and dyspnea due to exercise. This novel approach will have a significant impact on field, because it promises both additional insight into mechanisms of disease and immediate therapeutic options.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of IPF
* 40-85 years of age
* 6-minute walk distance 150-500 m
* FVC 40-90% predicted
* DLCO 30-90% predicted

Exclusion Criteria:

* Severe pulmonary hypertension
* Severe heart failure
* FEV1/FVC < 0.7

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-07; Primary Completion 2008-10 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Jackson, MD, Principal Investigator — VA Medical Center, Miami
Locations (1):
- VA Medical Center, Miami, Miami, Florida, United States

REFERENCES:
- [Result] Jackson RM, Glassberg MK, Ramos CF, Bejarano PA, Butrous G, Gomez-Marin O. Sildenafil therapy and exercise tolerance in idiopathic pulmonary fibrosis. Lung. 2010 Apr;188(2):115-23. doi: 10.1007/s00408-009-9209-8. Epub 2009 Dec 12. PMID 20012639
- [Result] Jackson R, Ramos C, Gupta C, Gomez-Marin O. Exercise decreases plasma antioxidant capacity and increases urinary isoprostanes of IPF patients. Respir Med. 2010 Dec;104(12):1919-28. doi: 10.1016/j.rmed.2010.07.021. Epub 2010 Aug 23. PMID 20739168

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2006-2009; U Miami and VA IPF clinics
Pre-assignment Details: Some were excluded after enrollment, because they did not meet entry criteria.
Groups:
- Sildenafil: Sildenafil 20 mg TID orally : Assessing the possible therapeutic benefit of sildenafil on exercise tolerance in IPF patients.
- Placebo: Control group: Identical Placebo 20 mg TID orally
Period: Overall Study
Arm/Group | Sildenafil | Placebo
Started | 14 | 15
Completed | 14 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sildenafil: Sildenafil 20 mg TID orally: Assessing the possible therapeutic benefit of sildenafil on exercise tolerance in IPF patients.
- Placebo: Identical Placebo: 20 mg TID orally
- Total: Total of all reporting groups
Arm/Group | Sildenafil | Placebo | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 11 | 13 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.9 (12.0) | 71.0 (6.2) | 70.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 11 | 12 | 23
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 29

OUTCOME MEASURES:

1. Secondary Outcome: Dyspnea Score (Borg Scale)
Description: The Dyspnea score or Borg Rating of Perceived Exertion (RPE) Scale score is a subjective rating of perceived exertion. In medicine this is used to document the patient's effort and exertion, breathlessness and fatigue during a physical test.
  The Dyspnea score ranges from 0 (No breathlessness at all) to 10 (Maximum or extremely strong breathlessness).
  IN this study the Specific Objective 2 was to assess and compare changes from baseline in pre- and post-exercise dyspnea in the sildenafil and placebo control groups.
Time Frame: 0 - 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sildenafil: Sildenafil 20 mg tid
  sildenafil: Assessing the possible therapeutic benefit of sildenafil on exercise tolerance in IPF patients.
- Placebo: Identical Placebo 20 mg tid
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 14 | 15
units on a scale
  Pre-Exercise Dypsnea score | 0.86 (1.77) | 0.38 (1.39)
  Post-Exercise Dypsnea score | 0.89 (2.11) | 0.15 (1.68)

2. Primary Outcome: Change in 6-minute Walk Test
Description: Distance in meters -- Distance (meters) walked in 6 minutes
Time Frame: 0 - 6 months
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Placebo: Identical Placebo 20mg tid orally
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 14 | 15
meters | -26 (45) | -7 (34)

ADVERSE EVENTS:
Time Frame: 3 years
Description: No additional follow up
Groups:
- Placebo: Control group
- Sildenafil: sildenafil : Assessing the possible therapeutic benefit of sildenafil on exercise tolerance in IPF patients.
Arm/Group | Placebo | Sildenafil
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 1/15 | 6/14
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=15) | Sildenafil (N=14)
Flushing (General disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Change in vision (Eye disorders) | 0 (0) | 1 (1)
Syncope (General disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No